CLINICAL TRIAL: NCT02698124
Title: Prospective Observation of the indUction Regimen for Acute Non-Promyelocytic Myeloid Leukemia in Elderly; Decitabine for Chemotherapy Unfit Korean Acute Myeloid Leukemia (AML) Patients in Real Practice
Brief Title: Decitabine for Chemotherapy Unfit Korean AML Patients in Real Practice
Acronym: PURPLE-D
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ulsan University Hospital (Other)
Collaborators: The Korean Society of Hematology, AML/MDS Working Party (Unknown)
Responsible Party: Principal Investigator, Hawk Kim, Professor, Ulsan University Hospital
Other Study IDs: AMLMDSWP-201601
Record Dates: First submitted 2016-02-19; First posted 2016-03-03 (Estimated); Last update posted 2016-03-07 (Estimated); Status verified 2016-03

CONDITIONS: Acute Myeloid Leukemia; Elderly; Intensive Chemotherapy Unfit
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Decitabine

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — miRNA, TET, whole genome sequencing
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Decitabine: Decitabine 20mg/m2 will be given IV daily on Days 1-5 in 28-day cycles. Treatment should be given for at least 4 cycles in the absence of unacceptable toxicity or disease progression requiring alternative therapy.
  Beyond 4 cycles, treatment should continue as long as the subject continues to benefit based on investigator's judgment of no definitive progression.
  Interventions: Drug: Decitabine

INTERVENTIONS:
Drug: Decitabine

SUMMARY:
Prospective multicenter, open-lab el, observational, single arm study of decitabine. Subjects will be elderly patients with newly diagnosed, treatment-naïve AML who are unfit to receive and not candidate for intensive induction chemotherapy (iIC)

ELIGIBILITY:
Inclusion Criteria:

1. Newly diagnosed and therapy-naïve AML (bone marrow or peripheral blood blast counts ≥20%)
2. 65 years of age or older
3. Taking informed consent with signature and date
4. Not eligible for iIC based on either:

i) ≥75 years of age ii) comorbidity iii) secondary AML iv) poor performance (ECOG ≥2) v) Poor-risk by NCCN Guideline version 1.2015 vi) subject's choice (refusal for iIC) investigator's judgement incompatible with iIC

Exclusion Criteria:

1. Candidate for iIC at the time of enrollment
2. Promyelocytic leukemia, or AML with t(15;17) or PML/RARα rearrangement
3. AML with t(9;22) or BCR/ABL rearrangement
4. Leukemia central nervous system involvement
5. Extramedullary myeloid sarcoma without bone marrow involvement
6. Prior treatment with decitabine or azacitidine of any cause
7. Any leukemia-specific therapy, except for hydroxyurea for reducing leukemic cells prior decitabine
8. Second malignancy currently requiring active therapy except breast or prostate cancer stable on or responding to endocrine therapy, or curatively resected non-melanoma skin cancer or intraepithelial cancer
9. Premenopausal woman
10. Severe active infection
11. Uncontrolled bleeding Hypersensitivity to decitabine

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: elderly patients with previously untreated AML who are ufit to receive and not considered candidates for iIC at the time of enrollment
Sampling Method: Probability Sample
Enrollment: 136 (Estimated)
Dates: Start 2016-03; Primary Completion 2019-08 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
The rate of complete remission | after 4 cycles of decitabine treatment (about 4 months)
  The rate of complete remission and complete remission with incomplete platelet recovery (CRp) will be measured by 4 cycles of decitabine treatment.

SECONDARY OUTCOMES:
The rate of composite CR | after 4 cycles of decitabine treatment (about 4 months)
  CR+CRp+ CR with incomplete blood count recovery (CRi)
Clinical benefit rate | after 4 cycles of decitabine treatment (about 4 months)
  cCR(CR+CRp+CRi)+ partial remission (PR)+ stable disease (SD)
Change of quality of life scale using EQ-5D-3L | after 4 cycles of decitabine treatment (about 4 months)
  Quality of life measurement by EQ-5D will be compared between pre- and post-decitabine therapy.
Change of quality of life scale using EORTC QLQ-C30 | after 4 cycles of decitabine treatment (about 4 months)
  Quality of life measurement by EORTC QLQ-C30 will be compared between pre- and post-decitabine therapy.
Number of participants with treatment-related adverse events as assessed by CTCAE v4.03 | until 4 cycles of decitabine treatment (about 4 months)
  CTCAE version 4.03

CONTACTS AND LOCATIONS:
Locations (1):
- Ulsan University Hospital, Ulsan, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kantarjian HM, Thomas XG, Dmoszynska A, Wierzbowska A, Mazur G, Mayer J, Gau JP, Chou WC, Buckstein R, Cermak J, Kuo CY, Oriol A, Ravandi F, Faderl S, Delaunay J, Lysak D, Minden M, Arthur C. Multicenter, randomized, open-label, phase III trial of decitabine versus patient choice, with physician advice, of either supportive care or low-dose cytarabine for the treatment of older patients with newly diagnosed acute myeloid leukemia. J Clin Oncol. 2012 Jul 20;30(21):2670-7. doi: 10.1200/JCO.2011.38.9429. Epub 2012 Jun 11. PMID 22689805
- [Result] Blum W, Garzon R, Klisovic RB, Schwind S, Walker A, Geyer S, Liu S, Havelange V, Becker H, Schaaf L, Mickle J, Devine H, Kefauver C, Devine SM, Chan KK, Heerema NA, Bloomfield CD, Grever MR, Byrd JC, Villalona-Calero M, Croce CM, Marcucci G. Clinical response and miR-29b predictive significance in older AML patients treated with a 10-day schedule of decitabine. Proc Natl Acad Sci U S A. 2010 Apr 20;107(16):7473-8. doi: 10.1073/pnas.1002650107. Epub 2010 Apr 5. PMID 20368434
- [Result] Mims A, Walker AR, Huang X, Sun J, Wang H, Santhanam R, Dorrance AM, Walker C, Hoellerbauer P, Tarighat SS, Chan KK, Klisovic RB, Perrotti D, Caligiuri MA, Byrd JC, Chen CS, James Lee L, Jacob S, Mrozek K, Bloomfield CD, Blum W, Garzon R, Schwind S, Marcucci G. Increased anti-leukemic activity of decitabine via AR-42-induced upregulation of miR-29b: a novel epigenetic-targeting approach in acute myeloid leukemia. Leukemia. 2013 Apr;27(4):871-8. doi: 10.1038/leu.2012.342. Epub 2012 Nov 26. PMID 23178755
- [Result] Suzuki H, Maruyama R, Yamamoto E, Kai M. DNA methylation and microRNA dysregulation in cancer. Mol Oncol. 2012 Dec;6(6):567-78. doi: 10.1016/j.molonc.2012.07.007. Epub 2012 Aug 10. PMID 22902148
- [Result] Kim Y, Cheong JW, Kim YK, Eom JI, Jeung HK, Kim SJ, Hwang D, Kim JS, Kim HJ, Min YH. Serum microRNA-21 as a potential biomarker for response to hypomethylating agents in myelodysplastic syndromes. PLoS One. 2014 Feb 4;9(2):e86933. doi: 10.1371/journal.pone.0086933. eCollection 2014. PMID 24503739
- [Result] Castoro RJ, Dekmezian M, Saraf AJ, Watanabe Y, Chung W, Adhab SE, et al. MicroRNA 124 and Its Role in Response to Epigenetic Therapy in Patients with Acute Mylogenous Leukemia and Myelodysplastic Syndrome. American Society of Hematology 2008; Abstract No. 598
- [Result] Cheson BD, Bennett JM, Kopecky KJ, Buchner T, Willman CL, Estey EH, Schiffer CA, Doehner H, Tallman MS, Lister TA, Lo-Coco F, Willemze R, Biondi A, Hiddemann W, Larson RA, Lowenberg B, Sanz MA, Head DR, Ohno R, Bloomfield CD; International Working Group for Diagnosis, Standardization of Response Criteria, Treatment Outcomes, and Reporting Standards for Therapeutic Trials in Acute Myeloid Leukemia. Revised recommendations of the International Working Group for Diagnosis, Standardization of Response Criteria, Treatment Outcomes, and Reporting Standards for Therapeutic Trials in Acute Myeloid Leukemia. J Clin Oncol. 2003 Dec 15;21(24):4642-9. doi: 10.1200/JCO.2003.04.036. PMID 14673054